CLINICAL TRIAL: NCT03746977
Title: Effects of Whole-body Electromyostimulation (WB-EMS), Physical Activity and Protein Supplementation on Lean Body Mass Maintenance During Caloric Restriction and Physical Activity Induced Weight Loss. A Randomized Controlled Study
Brief Title: Effects of WB-EMS and Protein Supplementation on LBM Maintenance During Intended Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Professor Dr. Wolfgang Kemmler, Principal Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WREPP
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Overweight; Obesity; Abdominal Obesity
Keywords: exercise; electromyostimulation; protein; weight reduction
MeSH Terms: conditions — Overweight; Obesity; Obesity, Abdominal; Motor Activity; Weight Loss | interventions — Proteins; Walking

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel group design with 3 study arms
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors were not aware of the status of the participants and were not allowed to ask correspondingly. Each of the participants were blinded according to the treatment and intervention. Participants of the three study groups were not in contact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- energy restriction and protein supplementation (Active Comparator): Energy restriction of 500 kcal/d and total Protein Uptake (including Supplementation) of 1.2 g/kg body mass/d
  Interventions: Dietary Supplement: Protein
- Energy restriction, walking and protein (Active Comparator): Energy restriction of 250 kcal/d, increased energy consumption by walking (250 kcal/d) and total protein uptake (including supplementation) of 1.5 g/kg body mass/d
  Interventions: Dietary Supplement: Protein; Behavioral: Walking
- Energy restriction, walking, protein and WB-EMS (Active Comparator): Energy restriction of 250 kcal/d, increased energy consumption by walking (250 kcal/d), total protein uptake (including supplementation) of 1.5 g/kg body mass/d and WB-EMS application 1,5x 20 min/week
  Interventions: Dietary Supplement: Protein; Behavioral: Walking; Behavioral: WB-EMS application

INTERVENTIONS:
Dietary Supplement: Protein — Protein supplementation 1.2 or 1.5 g/kg body mass/d
Behavioral: Walking — Walking with a volume corresponding to 250 kcal/d
  Arms: Energy restriction, walking and protein; Energy restriction, walking, protein and WB-EMS
Behavioral: WB-EMS application — WB-EMS application 1.5x 20 min/week
  Arms: Energy restriction, walking, protein and WB-EMS

SUMMARY:
The present study aimed to determine the effect of different interventions on lean body mass maintenance under weight loss conditions in overweight and obese premenopausal women. Three study groups were implemented: (1) Protein supplementation (only) group (2) Protein supplementation and walking intervention (3) Protein supplementation, walking and WB-EMS-application. All protocols were applied for 16 week of intervention.

A energy deficit of 500 kcal/d was intended however while group (1) focus consistently on energy restriction (500 kcal/d), in group (2) and (3) a combined physical activity (i.e. walking with a volume representing 250 kcal/d) and energy restriction (250 kcal/d) protocol was applied. Total protein uptake including protein supplementation was calculated to average around 1.2 g/kg body mass per day in groups (1) and 1.5 g/kg body mass/d in group (2) and (3). WB-EMS was applied 1.5x 20 min/week (i.e. each Tuesday and every second Thursday).

Primary study endpoint was LBM as determined by Dual Energy x-Ray Absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women 25-50 years old
* overweight/obesity (body fat rate equal or higher 30%)

Exclusion Criteria:

* medication and diseases affecting muscle and fat metabolism
* pregnant or parturition < 6 months
* any condition or medication that prevent proper physical activity or WB-EMS application
* holidays equal or more than 1 week during the intervention period
* other interventions with impact on the primary and core secondary outcome (i.e. body fat parameters) started during the last year.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Lean body mass | changes from baseline to 16 week follow-up
  Fat and bone free total body mass in kg

SECONDARY OUTCOMES:
Total Body Fat | changes from baseline to 16 week follow-up
  Total Body Fat in kg
Total Body Fat Rate | changes from baseline to 16 week follow-up
  Percent Total Body Fat Rate
Appendicular Skeletal Muscle Mass | changes from baseline to 16 week follow-up
  Lean Body Mass of the upper and lower limbs in kg
Visceral Body Fat | changes from baseline to 16 week follow-up
  Total visceral body fat in kg
Trunk fat | changes from baseline to 16 week follow-up
  Total trunk fat in kg
Metabolic Syndrome Z-Score | changes from baseline to 16 week follow-up
  Summarized Z-Score that included Z-Scores of blood lipids, lipoproteins, glucose, resting blood pressure and waist circumference. Cut-offs based on the definition of the International Diabetes Federations

CONTACTS AND LOCATIONS:
Overall Officials: Simon von Stengel, PhD, Study Chair — Institute of Medical Physics, FAU Erlangen-Nürnberg, Germany
Locations (1):
- Institute of Medical Physics University of Erlangen-Nurnberg, Erlangen, Germany